CLINICAL TRIAL: NCT07050914
Title: Comparison of McGrath Laryngoscope With Macintosh Laryngoscope in Obstetric Patients Undergoing Cesarean Section With Regards to Time of Intubation and Laryngeal View: A Randomized Controlled Trial
Brief Title: Comparison of McGrath Laryngoscope With Macintosh Laryngoscope in Obstetric Patients Undergoing Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sobia Khan, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-6490-20096
Record Dates: First submitted 2025-06-12; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group McGrath Laryngoscope (Experimental)
  Interventions: Device: McGrath Video Laryngoscope
- Group Macintosh Laryngoscope (Active Comparator)
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: McGrath Video Laryngoscope — A video laryngoscope.
  Arms: Group McGrath Laryngoscope
Device: Macintosh Laryngoscope — A classic laryngoscope.
  Arms: Group Macintosh Laryngoscope

SUMMARY:
The goal of this clinical trial is to compare the McGrath video laryngoscope with the Macintosh laryngoscope in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 45 years
* American society of Anesthesiologists (ASA) II patients

Exclusion Criteria:

* Category 1 Cesarean section
* Anticipated difficult airway
* Renal, hepatic, neuro-muscular, or cardiovascular illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Intubation time | 30 - 60 seconds from laryngoscope insertion in the oral cavity till detection of end tidal carbon dioxide trace.
Cormack Lehane grade | During laryngoscopy.
Pogo score | During laryngoscopy.

SECONDARY OUTCOMES:
Mean Arterial Blood Pressure | Before intubation and 1 minute after intubation
Heart Rate | Before intubation and 1 minute after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Khan, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yumul R, Elvir-Lazo OL, White PF, Sloninsky A, Kaplan M, Kariger R, Naruse R, Parker N, Pham C, Zhang X, Wender RH. Comparison of three video laryngoscopy devices to direct laryngoscopy for intubating obese patients: a randomized controlled trial. J Clin Anesth. 2016 Jun;31:71-7. doi: 10.1016/j.jclinane.2015.12.042. Epub 2016 Mar 23. PMID 27185681
- [Background] Arici S, Karaman S, Dogru S, Karaman T, Tapar H, Ozsoy AZ, Kaya Z, Suren' M. The McGrath Series 5 video laryngoscope versus the Macintosh laryngoscope: a randomized trial in obstetric patients. Turk J Med Sci. 2014;44(3):387-92. doi: 10.3906/sag-1306-71. PMID 25558638